CLINICAL TRIAL: NCT01102881
Title: Laxation and Satiety Response of Novel Dietary Fibers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Tate and Lyle Ingredients France (Industry); General Mills (Industry)
Responsible Party: Joanne Slavin, University of Minnesota
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 0902M60241
Record Dates: First submitted 2010-03-23; First posted 2010-04-13 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy adults

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- No fiber (Placebo Comparator): No fiber added to muffins or cereal
  Interventions: Dietary Supplement: placebo
- Fiber made from corn starch (Experimental): Muffins and cereal made with novel corn fiber
  Interventions: Dietary Supplement: Fiber made from corn starch
- Glucose polymer fiber (Experimental): Muffins and cereal made from glucose polymer fiber
  Interventions: Dietary Supplement: Glucose polymer fiber

INTERVENTIONS:
Dietary Supplement: Glucose polymer fiber — 20 grams of fiber per day split into two 10 gram doses administered as a breakfast cereal and a muffin or no-fiber breakfast cereal and muffin
  Arms: Glucose polymer fiber
Dietary Supplement: Fiber made from corn starch — 20 grams of fiber per day split into two 10 gram doses administered as a breakfast cereal and a muffin or no-fiber breakfast cereal and muffin
  Other Names: Dietary fiber made from corn starch
  Arms: Fiber made from corn starch
Dietary Supplement: placebo — low fiber breakfast cereal and muffin
  Arms: No fiber

SUMMARY:
Dietary fibers have previously been shown to affect laxation and satiety. Due to differences in structure and physical properties of dietary fibers, these effects may not be consistent across all fibers. Therefore as new dietary fibers are created or discovered the laxative and satiating effects should be investigated in order to verify these effects.

DETAILED DESCRIPTION:
This study was designed to test the laxative effects of two fibers a resistant starch made from corn and a glucose polymer fiber. The secondary aim of this study was to examine the satieting effects of these fibers. This trial was double-blind and placebo controlled. On the first day of the study subjects consumed the breakfast cereal and milk and were instructed to complete visual analog scales periodically to test acute satiety. Subjects also completed diet records and tolerance questionnaires on days 1,2, and 10. Additionally subjects completed another satiety survey on day 10 to test chronic satiety. Whole gut transit time, fecal weight, and fecal chemistry was tested by swallowing radioopaque pellets on day 6 and collecting every fecal sample for the 5 days thereafter.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age 18-65
* non-smoking
* not taking medication
* non-dieting (weight stable in prior 3 months)
* BMI 18-30
* English literacy

Exclusion Criteria:

* do not regularly consume breakfast
* food allergies to ingredients found in study product
* dislike of cereal or muffins
* BMI <18 or >30
* diagnosed with cardiovascular, renal, or hepatic disease
* diabetes mellitus (fasting blood glucose > 126 mg/ml)
* cancer in previous 5 years (except basal cell carcinoma of the skin)
* any gastrointestinal disease or condition
* recent bacterial infection (< 3 months)
* recent or concurrent participation in an intervention research study
* history of drug or alcohol abuse in prior 6 months
* use of lipid-lowering, anti-hypertensive, or anti-inflammatory steroid medications vegetarians people who eat more than approximately 15 grams of dietary fiber per day women who are pregnant or lactating women with irregular menstrual cycles consumption of prebiotics or probiotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time determined by radio-opaque pellets | 5 day fecal collection
  Determine whole gut transit time by x-raying fecal samples after swallowing radio-opaque pellets

SECONDARY OUTCOMES:
Satiety | 0, 15, 30, 45, 60, 90, 120, 180, 240 minutes postprandially
  Measure hunger, fullness, satisfaction, and prospective food consumption using a 100 mm line
Breath Hydrogen concentration after consumption of test cereal | 0 and 240 minutes postprandially
  Subjects expel air into a storage bag, which is then injected into a gas chromatograph and determine the hydrogen concentration. Hydrogen gas is an indicator of fermentation in the large intestine.
Ad libitum food intake | 24 hours, 48 hours, and 10 days after the start of treatment
  24 hour food diary
Gastrointestinal Tolerance | 24 hours, 48 hours, and 10 days after the start of the treatment
  Rank severity of flatuence, bloating, abdominal cramps, stomach noises, nausea, diarrhea, and constipation on a 10 point scale.
Fecal chemistry | 6-10 days after the start of treatments
  Determination of fecal pH and short-chain fatty acid concentration

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States